CLINICAL TRIAL: NCT02643563
Title: Comparison of the Analgesic Duration of 0.5% Bupivacaine With 1:200,000 Epinephrine Versus 0.5% Ropivicaine Versus 1 % Ropivicaine for Low Volume Ultrasound-guided Interscalene Brachial Plexus Block
Brief Title: Analgesic Duration of Long Acting Local Anesthetics for Low Volume Ultrasound-guided Interscalene Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Ben Safa, Anesthesiologist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 456-2014
Record Dates: First submitted 2015-12-26; First posted 2015-12-31 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Brachial Plexus Block; Anesthetics, Local
Keywords: Brachial Plexus Block; Anesthetics, Local
MeSH Terms: interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ropivacaine 0.5% (Experimental): Low volume (5 ml) Interscalene Block with Ropivacaine 0.5%
  Interventions: Drug: Ropivacaine 0.5%
- Ropivacaine 1% (Active Comparator): Low volume (5 ml) Interscalene Block with Ropivacaine 1%
  Interventions: Drug: Ropivacaine 1%
- Bupivacaine 0.5% + epinephrine 1:200,000 (Active Comparator): Low volume (5 ml) Interscalene Block with Bupivacaine 0.5% + epinephrine 1:200,000
  Interventions: Drug: Bupivacaine 0.5% + epinephrine 1:200,000

INTERVENTIONS:
Drug: Ropivacaine 0.5% — Ropivacaine 0.5% is used for low-volume ultrasound-guided interscalene brachial plexus block.
  Arms: Ropivacaine 0.5%
Drug: Ropivacaine 1% — Ropivicaine 1% is used for low-volume ultrasound-guided interscalene brachial plexus block.
  Arms: Ropivacaine 1%
Drug: Bupivacaine 0.5% + epinephrine 1:200,000 — Bupivacaine 0.5% + epinephrine 1:200,000 is used for low-volume ultrasound-guided interscalene brachial plexus block.
  Arms: Bupivacaine 0.5% + epinephrine 1:200,000

SUMMARY:
Severe pain following shoulder surgery is common and remains a major challenge. The interscalene nerve block is well suited for operations on the shoulder or upper arm, for providing surgical anesthesia as well as prolonged effective postoperative analgesia.

Modern ultrasound guided ISB (US-ISB) allows for more accurate, targeted deposition of local anesthetic. The current trend is to lower the volume of local anesthetic for ultrasound-guided interscalene block in order to reduce potential complications such as phrenic nerve paralysis and local anesthetic toxicity. However, at low volumes the analgesic duration of the block could be compromised. Studies to elucidate the best local anesthetic agent, concentration and adjuncts to prolong analgesia at low volumes are needed. Ropivacaine and Bupivacaine are long acting local anesthetics commonly used for peripheral nerve blocks, however, there are no studies comparing their analgesic duration in the setting of low volume interscalene block to date.

This study will investigate the analgesic duration of 0.5% Ropivacaine versus 0.5% Bupivacaine with 1:200,000 epinephrine versus 1% Ropivacaine for low volume US-ISB.

This study aims to conduct a comparison of the duration of post operative analgesia achieved by these agents, hence allowing the appropriate local anesthetic agent and concentration selection in low-volume techniques.

DETAILED DESCRIPTION:
Hypothesis:

0.5 % Bupivacaine with 1:200,000 epinephrine and 1% Ropivicaine provide longer duration analgesia than 0.5% Ropivicaine following a low dose ultrasound guided interscalene brachial plexus block (US-ISB)

Background and Rationale:

Severe pain following shoulder surgery is common and remains a major challenge. The interscalene approach to the brachial plexus is particularly well suited for operations on the shoulder or upper arm for providing surgical anesthesia as well as prolonged effective postoperative analgesia.

Despite the benefits, the interscalene approach may present risks and complications. Common complications of the interscalene nerve block include phrenic nerve blockade , Horner's syndrome, recurrent laryngeal nerve blockade, and vasculature puncture. Rare, but potentially devastating, complications include carotid artery puncture and intervertebral artery injection, pneumothorax, subdural injection, intervertebral foramina injection resulting in spinal or epidural anesthesia, nerve injury and local anesthetic toxicity have been reported.

The use of ultrasound (US) in regional anesthesia has allowed for easy visualization of the nerve, the needle, and the dispersion of the anesthetic, facilitating adequate injection in the perineural region. US-guided blocks have been associated with high success rates, reduced latencies, and reduced LA doses. A number of recent studies have confirmed that the use of ultrasound (US) also allows for a significant reduction in the local anesthetic volume for an effective interscalene nerve block. This reduction in volume of local anesthetic not only translates into reduced risk of local anesthetic toxicity but also a substantial reduction in the incidence of phrenic nerve paralysis.

Based on the available research to date it appears that an effective interscalene block can be performed with a small volume of 5 ml of local anesthetic while minimizing the incidence of phrenic nerve palsy and local anesthetic toxicity. Based on the limited data available thus far the analgesic duration of the block does not appear to be compromised with the low volume techniques. However the critics of the low volume US-ISB persist with the belief that low-volume techniques, with their reduced local anesthetic dose, inherently produce a shorter duration block of lesser quality compared to higher volume. To date there are no studies comparing the analgesic duration of available and commonly used long acting local anesthetics in the setting of low-volume ISB technique.

Bupivacaine and ropivicaine are the preferred long acting local anesthetics as they provide prolonged analgesia in the postoperative period. However, ropivacaine due to its reduced lipophilicity is generally considered less potent than bupivacaine with a shorter duration of action . The magnitude of this potency difference however is not clearly quantified and differs with varying techniques. In some studies, the potency difference amounts up to 50% whereas in other studies the difference is negligible. This may be due to the fact that this potency difference is dose dependent phenomenon. Ropivacaine has similar potency to bupivacaine at higher doses (e.g., doses required for peripheral nerve blocks for surgical anesthesia), ropivacaine is less potent than bupivacaine at lower doses, such as those used for epidural or intrathecal analgesia .

Clearly for low volume US-ISB, ropivicaine's potentially improved safety profile becomes clinically insignificant, and the dose dependent reduced potency may play an important role in decreasing the duration of analgesia. Previous studies looking at the performance of ropivicaine and bupivicaine for upper extremity peripheral nerve blocks have only been done in high volume settings. In these studies the high dose of local anesthetic used may have masked any difference in potency of bupivacaine and ropivicaine.

Clearly future studies are needed to better define the analgesic duration of low volumes US-ISB and determine the effects of different local anesthetics, different concentrations and adjuncts on the duration and quality of the block at these low volumes.

Specific Objective

To investigate the analgesic duration of 0.5% ropivacaine versus 0.5% bupivacaine with 1:200,000 epinephrine versus 1% ropivacaine for low volume US-ISB.

Protocol:

Patients scheduled for arthroscopic shoulder surgery will be approached for participation by research assistants in the pre-operative anesthetic clinic. Patients providing informed consent will be allocated to one of three groups using a computer generated random number table and blinding of group allocation will be maintained with sequentially numbered, sealed, opaque envelopes.

On the day of surgery, patients will be pre-medicated with oral acetaminophen 1000mg (650mg if < 60kg), and oral celecoxib 400mg (200mg if < 60kg). Once intravenous access is secure and standard monitors applied (electrocardiogram, non-invasive blood pressure cuff, continuous oxygen saturation), patients will receive sedation with intravenous midazolam (1-2mg). The lateral aspect of the neck including the supraclavicular fossa ipsilateral to the surgical site will be cleansed with an isopropyl alcohol/chlorhexidine gluconate solution. The US-guided ISB will be performed under sterile conditions by a staff regional anesthesiologist, or regional anesthesia fellow. The ISB will be performed using a 13-6 MHz 38-mm linear US probe with appropriate sterile barrier (M-Turbo®; SonoSite Inc., Bothell, WA) at the upper trunk level via posterior approach with a 22-gauge insulated 50-mm regional block needle (Stimuplex®; B.Braun Medical, Bethlehem, PA). After satisfactory position of the needle tip is achieved and visualized, the injectate will be administered slowly.

The local anesthetic injectate will be prepared in a blinded syringe by trained anesthesia assistants that are aware of group allocation but will take no further part in study procedures or assessments. This individual will prepare the injectate in a 5ml syringe.

All other personnel - patients, anesthesiologists performing the ISB or caring for the patient in the operating theatre, surgeons, research assistants performing outcome measures, and statisticians - will remain blinded.

The block will be assessed at 20 minute intervals, using loss of pinprick sensation to C5/C6 dermatome and strength of shoulder abduction. Patients will be excluded if there is no evidence of both sensory and motor block at 20 minutes.

Patients will undergo general anesthesia with a standardized induction technique using fentanyl 1mcg/kg, and propofol 1-3mg /kg. Endotracheal intubation will be facilitated with rocuronium 0.6mg/kg if necessary or a laryngeal mask airway can be placed for spontaneously breathing patients. Anesthesia will be maintained using the inhalational anesthetic sevoflurane (Abbott Corp) with an end-tidal concentration of 1.4 - 2%. Muscle relaxation will be reversed using a combination of neostigmine (0.04mg/kg) and glycopyrrolate (0.007mg/kg) in necessary. Supplementary intraoperative opioids for pain (systolic blood pressure or heart rate increase from baseline of greater than 10% from surgical stimulus) will be given at the discretion of the attending anesthesiologist (intravenous hydromorphone [0.2 mg per bolus] or fentanyl [25 ug per bolus]) intravenous . Standard anti-emetic prophylaxis with the serotonin antagonist ondansetron will be given.

Upon arrival to the recovery room, pain (Verbal Response Score ≥4 or patient request for analgesia) will be treated with hydromorphone in 0.2-0.4mg increments every 5 minutes as needed. Once oral intake is initiated, patients will receive one of two oral analgesic preparations as needed: Tylenol #3® (acetaminophen 325 mg/codeine 30 mg/caffeine 15 mg per tablet), or oxycocet (acetaminophen 325 mg/oxycodone HCl 5 mg per tablet) if intolerant to codeine. Upon discharge from hospital, patients will receive a prescription for Tylenol #3® as needed, or oxycocet if intolerant to codeine. After discharge, patients will complete a home diary and return to the study team using a stamped, return-addressed envelope. Patients will be asked to record the time at which they first experience pain at the surgical site, the time when they first consume prescribed opioid analgesics for surgical site pain and regain normal (or baseline equivalent) strength in their biceps and hand. On postoperative days (POD) 1, 2 at 12h00 patients will be requested to document interval oral analgesic consumption, presence of nausea or vomiting, presence of weakness in the operative arm, and presence of paresthesia (numbness or tingling) in the operative arm. The doses of oral codeine or oxycodone consumed by each patient will be converted into equianalgesic doses of conversion ratios will be employed according to the general monograph for opioids in the Canadian Pharmacists' Association Compendium of Pharmaceuticals and Specialties (36th ed., 2001) as follows: oral oxycodone: oral morphine sulphate = 1:2, and oral codeine: oral morphine sulphate = 6.6:1.

Sample size calculation

Based on the investigator's clinical experience with low dose US-ISB (Ropivacaine 0.5% 5ml) as well as previously published work, Investigators expect analgesic duration of 12 hours with a standard deviation of 4 hours. The sample size calculation is based on being able to detect a difference of 30% (3.6 hours ) in duration of analgesia between the three groups.

It is estimated that 57 patients are required (19 per group) to achieve 80% power to detect differences among the means versus the alternative of equal means using an F test with a 0.05 significance level. The size of the variation in the means is represented by their standard deviation, which is 1.70. The common standard deviation within a group is assumed to be 4.00. To account for incomplete data or loss to follow-up, the plan is to recruit 60 patients total.

Data collection

Data will be collected on a customized case report form that includes all relevant demographic and intra-operative data as well as each outcome sought. Patients will be provided with a home diary to complete that will capture all outcomes sought that are not obtained in hospital.

Statistical analysis

Demographic data will be summarized and expressed using appropriate measures of central tendency and dispersion for continuous data, and frequency for categorical data. The primary outcome, time to first sensation of pain at the surgical site, will be summarized as mean (SD) or median (IQR) after testing the data for normality with the Kolmogrov Smirnoff test. This will also determine whether groups will be compared with the t-test (for normally distributed data) or Kaplan Meier Survival Curves (for skewed data). Secondary outcomes that are time based will also be assessed in the above manner (time to first analgesic request, duration of motor block). Continuous secondary outcomes (opioid consumption, VRS, room air SpO2) will be assessed with repeated measures ANOVA or the Mann Whitney U-test for non-parametric data. Categorical outcomes will be compared with the Chi square or Fisher's exact test as necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing arthroscopic shoulder surgery at Sunnybrook Health Sciences Centre
2. ASA functional status class I to III
3. BMI < 35 kg/m2

Exclusion Criteria:

1. Lack of patient consent
2. Allergy to bupivacaine or ropivacaine
3. BMI > 35 kg/m2
4. Contraindications to ISB including severe Chronic Obstructive Pulmonary Disease (Forced expiratory volume < 40% predicted), coagulopathy, pre-existing neurologic deficit in ipsilateral upper extremity, localized infection
5. Pregnant or nursing females
6. Chronic opioid use defined as > 30mg oral morphine equivalent per day

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2019-03 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Duration of analgesic block | 48 hours
  Defined as time from end of injection to first sensation of pain at surgical site

SECONDARY OUTCOMES:
Time to first opioid consumption | 24 hours or less
  Defined as time from end of injection to time to oral opioid consumption
Duration of motor block | 24 hours or less
  Defined as time from end of injection to time of preoperative biceps and hand strength
Diaphragmatic dysfunction assessed by ultrasound | 4 hours
  Assessed at at 4 hours post block compared to pre-operative values
Opioid consumption | 24 and 48 hours
  Cumulative opioid consumption at 24 and 48 hours
Pain VAS scores | 4, 8, 12, 24, 48 hours
  Pain VAS scores at 4, 8, 12, 24, 48 hours (patient diary)
Vital capacity | 4 hours
  Assessed at at 4 hours post block compared to pre-operative values

CONTACTS AND LOCATIONS:
Overall Officials: Ben Safa, MD, Principal Investigator — Sunnybrook Health Sciences Center
Locations (1):
- Holland Orthopedic and Arthritic Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Safa B, Flynn B, McHardy PG, Kiss A, Haslam L, Henry PD, Kaustov L, Choi S. Comparison of the Analgesic Duration of 0.5% Bupivacaine With 1:200,000 Epinephrine Versus 0.5% Ropivacaine Versus 1% Ropivacaine for Low-Volume Ultrasound-Guided Interscalene Brachial Plexus Block: A Randomized Controlled Trial. Anesth Analg. 2021 Apr 1;132(4):1129-1137. doi: 10.1213/ANE.0000000000005373. PMID 33464760